CLINICAL TRIAL: NCT04269369
Title: Implementation of Pre-emptive Geno- and Phenotyping in 5-Fluorouracil- or Capecitabine-treated Patients With the Aim of Reducing Toxicity
Brief Title: Implementation of Pre-emptive Geno- and Phenotyping in 5-Fluorouracil- or Capecitabine-treated Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FluorouracilCapecitabine001
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Colon Cancer; Stomach Tumor; Anal Tumor; Pancreas Cancer; Esophageal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Stomach Neoplasms; Anus Neoplasms; Pancreatic Neoplasms; Esophageal Neoplasms | interventions — Fluorouracil

STUDY DESIGN:
Intervention Model Description: In a subgroup of patients, a parallel study model will be used. In the group of patients with genotype "wild type" and phenotype "intermediate metabolizer", a comparison will be made between group A with dosage according to French guidelines and group B with dosage according to literature. After obtaining written informed consent, patients will be randomized in a 1:1 ratio to one of the two study groups.
Masking Description: The study is not blinded (not for the patients participating in the trial and not for the treating physicians).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Dosage according to French guidelines
  Interventions: Drug: 5-Fluorouracil
- Group B (Experimental): Dosage according to literature
  Interventions: Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: 5-Fluorouracil — The aim of this study is to investigate if the systematic implementation of pre-emptive geno- and phenotyping, and therefore a dose reduction based on the French guidelines and the literature during the first month of treatment, reduces grade 3 or greater toxicity in patients treated with 5-FU or capecitabine. Therefore a dosing table was obtained by combining the results of the study by Henricks et al., Launay et al. and Yang et al. and the recommendations from the French HAS guideline. The treatment schedule then will be discussed by the team of doctors and paramedics at the weekly MOC (multidisciplinary cancer consultation). Complementary, the pharmacist provides dose advice with regard to the start of 5-FU or capecitabine treatment.
  In a subgroup, the group of patients with genotype "wild type" and phenotype "intermediate metabolizer", a comparison will be made between group A with dosage according to French guidelines and group B with dosage according to literature.

SUMMARY:
The aim of this study is to investigate if the systematic implementation of pre-emptive geno- and phenotyping, and therefore a dose reduction based on the French guidelines and the literature during the first month of treatment, reduces grade 3 or greater toxicity in patients treated with 5-FU (5-fluorouracil) or capecitabine.

Therefore, a monocentric, partial prospective and partial retrospective trail was designed.

DETAILED DESCRIPTION:
5-FU (5-fluorouracil) and its oral prodrug capecitabine are commonly used drugs in various chemotherapy regimens. According to the literature, approximately 30% of the patients experience at least a grade three toxicity during treatment, mainly characterized by diarrhea, mucositis, hematological toxicity or hand-foot syndrome. This toxicity can lead to discontinuation or interruption of the therapy, hospitalization and in 1% of the cases even to mortality. This leads to an increase in health care costs, mainly driven by the cost of hospitalization.

The metabolism of 5-FU and its prodrug is primarily determined by the dehydropyrimidine dehydrogenase (DPD) enzyme. The gene encoding for this enzyme, the DPYD, is known for his genetic polymorphism. Five percent of the population has a partial DPYD deficiency and 0.01 to 0.1 percent has a full DPYP deficiency. Partial deficiency leads to a reduced activity of DPD and therefore to a reduced degradation of 5-FU or capecitabine to its inactive metabolites. This leads to an increased toxicity. The four DPYD variants considered most clinically relevant are DPYD * 2A, DPYD * 13, c.1236G> A and c.2846A> T. Patients with polymorphisms DPYD * 2A and DPYD * 13 have no residual enzyme activity, while in patients with polymorphisms 1236G> A and c.2846A> T, there is still partial enzyme activity present. In addition to genotyping, partial DPYD deficiency can also be detected by phenotyping. In the case of reduced enzyme activity of DPYD, the degradation of uracil is disturbed, causing an increase in uracil and a decrease in UH2 in plasma. There is a strong correlation between the UH2 / U ratio in plasma and the halflife, clearance and plasma levels of 5-FU.

French guidelines, HAS (La Haute Autorité de santé), recommend to adjust the dose of these drugs at the start of treatment based on the results of both the genetic and phenotypic studies.

The aim of this study is to investigate if the systematic implementation of pre-emptive geno- and phenotyping, and therefore a dose reduction based on the French guidelines and the literature during the first month of treatment, reduces grade 3 or greater toxicity in patients treated with 5-FU or capecitabine.

Therefore, a monocentric, partial prospective and partial retrospective trail was designed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* WHO (world health organization) classification 0,1 or 2
* A suspected start with 5-FU or capecitabine in mono or combination therapy
* The knowledge of the result of the geno and phenotyping before the start of the treatment

Exclusion Criteria:

* Not meeting inclusion criteria
* Homozygote genotype or uracil 100 ng/ml or greater
* The lacking of the result of the geno and / or phenotyping before the start of treatment
* Patients who received 5-FU or capecitabine in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-02-18 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
The frequency of severe ﬂuoropyrimidine-related toxicity | about 3 months
  The primary endpoint of the study is the frequency of severe (National Cancer Institute Common Terminology Criteria for Adverse Events version 5 grade ≥3) ﬂuoropyrimidine-related toxicity across the entire treatment duration. Toxicity incidence between DPYD variant allele carriers and DPYD wild-type patients and poor or intermediate metabolizers and extensive metabolizers will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: An Lambaerts, Principal Investigator — Jessa Hospital

IPD SHARING:
Plan to Share IPD: No